CLINICAL TRIAL: NCT04503577
Title: Prospective Bladder Cancer Infrastructure: an Infrastructure for Observational and Interventional Bladder Cancer Research (ProBCI)
Brief Title: Prospective Bladder Cancer Infrastructure (ProBCI)
Acronym: ProBCI
Status: Recruiting | Type: Observational
Sponsor: Prospective Bladder Cancer Infrastructure Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ProBCI
Record Dates: First submitted 2020-08-04; First posted 2020-08-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Prospective cohort
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Bladder cancer patients

SUMMARY:
Prospective nation-wide cohort of high-risk non-muscle-invasive, muscle-invasive and metastatic bladder cancer in the Netherlands

ELIGIBILITY:
Inclusion Criteria:

* Bladder cancer
* Any stage except Ta
* 18 years or older
* Written informed consent

Exclusion Criteria:

* No exclusion criteria

Note: participation in ProBCI does not exclude the patient from participation in other studies.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Bladder cancer patients with high-risk non-muscle-invasive bladder cancer (T1, Tis or Ta+cis), muscle-invasvie bladder cancer (T2-4, any N, M0/X), and metastatic bladder cancer (any T, any N, M1a/b)
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 2020-10-04 (Actual); Primary Completion 2040-12-31 (Estimated); Study Completion 2041-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 10 years
  Alive/death/emigrated

SECONDARY OUTCOMES:
Progression-free survival | 10 yeas
  Progression/no progression
Recurrence-free survival | 10 yeas
  Recurrence/no recurrence
Health-related quality of life | 2 years
  EQ-5D (EuroQol-Five Dimensions)
Cancer-specific health-related quality of life | 2 years
  QLQ-C30 (Quality of Life Questionnaire-Cancer)

CONTACTS AND LOCATIONS:
Locations (23):
- Netherlands (23):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - ZGT, Almelo
  - Meander Medical Center, Amersfoort
  - Amsterdam UMC, location VUMC, Amsterdam
  - Rijnstate, Arnhem
  - Amphia Ziekenhuis, Breda
  - Albert Schweitzer Hospital, Dordrecht
  - Ziekenhuis Gelderse Vallei, Ede
  - Treant Hospital, Emmen
  - University Medical Center Groningen, Groningen
  - Spaarne Gasthuis, Hoofddorp
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Alrijne Ziekenhuis, Leiderdorp
  - Maastricht University Medical Center, Maastricht
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Radboud univerisity Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Zuyderland, Sittard
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
  - University Medical Center Utrecht, Utrecht
  - VieCuri, Venlo
  - SKB Winterswijk, Winterswijk
  - Isala, Zwolle

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data are available upon request to other research groups (please see www.probci.nl for procedure).
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: please see www.probci.nl for procedure
Access Criteria: please see www.probci.nl for procedure
URL: http://www.probci.nl

REFERENCES:
- [Derived] Richters A, Meijer RP, Mehra N, Boormans JL, van der Heijden AG, van der Heijden MS, Kiemeney LA, Aben KK. Prospective bladder cancer infrastructure for experimental and observational research on bladder cancer: study protocol for the 'trials within cohorts' study ProBCI. BMJ Open. 2021 May 18;11(5):e047256. doi: 10.1136/bmjopen-2020-047256. PMID 34006553
- [Derived] Richters A, Mehra N, Meijer RP, Boormans JL, van der Heijden AG, Smilde TJ, van der Heijden MS, Kiemeney LA, Aben KK. Utilization of systemic treatment for metastatic bladder cancer in everyday practice: Results of a nation-wide population-based cohort study. Cancer Treat Res Commun. 2020;25:100266. doi: 10.1016/j.ctarc.2020.100266. Epub 2020 Dec 8. PMID 33316557